CLINICAL TRIAL: NCT07022509
Title: Outcome Of Matrix Rotation Versus Single Incision Lateral Sulcus Mammoplasty In The Upper Quadrant Breast Carcinomas
Brief Title: Matrix Rotation Flap Versus Single Incision Lateral Sulcus Mammoplasty
Acronym: SLIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Osama Ragaa Abdelraouf Ibrahim, Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC 9-4-2022; PNURSP2025R168 (Other Grant/Funding Number: Princess Nourah bint Abdulrahman University)
Record Dates: First submitted 2025-05-30; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: breast cancer; Oncology; MRF; SLIM
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Statisticians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group MRF (Experimental): Matrix rotation flap MRF surgical procedure
  Interventions: Other: Technique surgery
- Group SLIM (Experimental): Single Incision Lateral Sulcus Mammoplasty (SLIM).
  Interventions: Other: proceduder surgery

INTERVENTIONS:
Other: proceduder surgery — The single-incision lateral sulcus mammoplasty is a breast-conserving surgical technique that involves making a single incision along the lateral aspect of the inframammary fold or within the natural skin crease of the lateral sulcus. This approach provides direct access to the lateral quadrants of the breast, which are commonly affected in breast carcinoma, allowing for effective tumor excision while preserving the breast contour.
  In SILSM, the incision is carefully planned to align with natural anatomical lines, ensuring optimal cosmetic results and minimal visible scarring. Through this lateral access point, the surgeon performs both tumor resection and glandular reshaping. The technique often involves mobilization and rearrangement of the remaining breast tissue to fill the defect left by the tumor excision, thereby maintaining breast symmetry and volume.
  This techn
  Arms: Group SLIM
Other: Technique surgery — The matrix rotation flap is a versatile oncoplastic surgical technique employed in the reconstruction of partial breast defects following tumor excision. This method involves the creation of a rotational skin and glandular flap, mobilized from adjacent breast tissue, typically using an inferolateral or inferomedial pedicle. The flap is designed in a curvilinear or semicircular fashion, allowing it to rotate into the defect site while maintaining adequate vascular supply.
  The MRF technique is particularly useful for defects in the lower quadrants of the breast, where direct tissue advancement may be limited. The surgeon carefully outlines a skin paddle adjacent to the resection cavity and undermines the surrounding breast parenchyma. The flap is then rotated and inset into the tumor bed to fill the defect, with the skin paddle contributing to both volume replacement and skin resurfacing if required.
  This approach provides robust coverage of the surgical cavity, helps restore breast co
  Arms: Group MRF

SUMMARY:
The study seeks to compare the single-incision lateral mammoplasty technique with the matrix rotation flap in patients with breast carcinoma. The primary outcome assessed is postoperative complications, while secondary outcomes include cosmetic appearance and patient satisfaction.

DETAILED DESCRIPTION:
This study is designed to conduct a comprehensive comparison between two breast-conserving surgical techniques used in the treatment of breast carcinoma: the single-incision lateral mammoplasty and the matrix rotation flap. These procedures are employed to achieve both oncologic safety and aesthetic preservation in patients undergoing surgery for breast cancer.

The primary objective of the study is to evaluate and compare the incidence and nature of postoperative complications associated with each technique. This includes, but is not limited to, wound healing issues, infection rates, hematoma or seroma formation, and any need for reoperation.

Secondary objectives focus on assessing the cosmetic outcomes and the overall satisfaction of the patients post-surgery. Cosmetic evaluation will be conducted through both surgeon-assessed and patient-reported outcomes, utilizing standardized scoring systems and photographic documentation. Patient satisfaction will be measured through validated questionnaires designed to capture perceptions of body image, aesthetic results, and quality of life following the procedure.

By systematically analyzing these parameters, the study aims to determine which technique offers a more favorable balance of surgical safety, aesthetic quality, and patient satisfaction, thereby guiding clinical decision-making in breast-conserving surgery for breast carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Upper Quadrant Breast Carcinomas.

Exclusion Criteria:

* Patients with T4 tumors, inflammatory breast cancer and distant metastasis, multi-centric breast cancer in more than one quadrant and diffuse microcalcifications were excluded from the study.

Ages: 42 Years to 61 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 4 weeks
  The total number (percentage) of participants in each group who got post-operative complications such as wound infection, hematoma, and seroma.

SECONDARY OUTCOMES:
Asthetic outcomes | 6 months
  Vancouver's scar scale with ranges from 0 (normal skin) to 13 (worst scar possible)
Patients' satisfaction | 6 months
  Five-point Likert scale with one being excellent, two good, three fair, four poor, and five bad. The higher the score, the worse is the result.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Benha University, Benha, Egypt, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Will be available upon approval of the funding institute

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- See also: pubmed official site — https://pubmed.ncbi.nlm.nih.gov/30620402/